CLINICAL TRIAL: NCT06516289
Title: Neoadjuvant Treatment of gBRCA-Mutated HER2-Negative Breast Cancer With HRS-1167 and Famitinib/ HRS-1167, Famitinib and Camrelizumab: A Prospective, Open-label, Multicenter, Phase II Trial
Brief Title: Neoadjuvant Treatment of gBRCA-Mutated HER2-Negative Breast Cancer With HRS-1167 and Famitinib ± Camrelizumab
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-N074
Record Dates: First submitted 2024-07-01; First posted 2024-07-23 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: BRCA-Mutated Breast Carcinoma; HER2-negative Breast Cancer
MeSH Terms: interventions — famitinib; camrelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Safety run-in (Experimental): HRS-1167 + famitinib
  Interventions: Drug: HRS-1167; Drug: Famitinib
- Phase 2: Cohort A (HR+/HER2-, gBRCAm) (Experimental): HRS-1167 + famitinib, RP2D
  Interventions: Drug: HRS-1167; Drug: Famitinib
- Phase 2: Cohort B (HR-/HER2-, gBRCAm) (Experimental): HRS-1167 + famitinib, RP2D
  Interventions: Drug: HRS-1167; Drug: Famitinib
- Phase 2: Cohort C (HR+/HER2-, gBRCAm expansion cohort) (Experimental): HRS-1167 + famitinib, (RP2D) + camrelizumab
  Interventions: Drug: HRS-1167; Drug: Famitinib; Drug: Camrelizumab
- Phase 2: Cohort D (HR-/HER2-, gBRCAm expansion cohort) (Experimental): HRS-1167 + famitinib, (RP2D) + camrelizumab
  Interventions: Drug: HRS-1167; Drug: Famitinib; Drug: Camrelizumab

INTERVENTIONS:
Drug: HRS-1167 — a highly selective PARP1 inhibitor
Drug: Famitinib — a tyrosine kinase inhibitor targeting VEGFR2, PDGFR, and c-kit
Drug: Camrelizumab — a humanised anti-programmed death-1 (anti PD-1) antibody
  Arms: Phase 2: Cohort C (HR+/HER2-, gBRCAm expansion cohort); Phase 2: Cohort D (HR-/HER2-, gBRCAm expansion cohort)

SUMMARY:
This study is a prospective, open-label, multi-center, phase II clinical trial designed for HER2-negative breast cancer with pathogenic mutations in the germline gene (gBRCA1/2) that were indicated for neoadjuvant chemotherapy. The characteristics of this study are a precision treatment scheme without chemotherapy, the scheme of HRS-1167 combined with famitinib neoadjuvant therapy for patients with gBRCA mutations is explored, and the efficacy of combined immunotherapy is further explored according to the efficacy of the combination of the two drugs.

DETAILED DESCRIPTION:
This study is a prospective, open-label, multi-center, phase II clinical trial designed for HER2-negative breast cancer with pathogenic mutations in the germline gene (gBRCA1/2) that were indicated for neoadjuvant chemotherapy. The characteristics of this study are a precision treatment scheme without chemotherapy, the scheme of HRS-1167 combined with famitinib neoadjuvant therapy for patients with gBRCA mutations is explored, and the efficacy of combined immunotherapy is further explored according to the efficacy of the combination of the two drugs. The study consists of a safety run-in period to explore the safety of HRS-1167 combined with famitinib, which is used to provide a recommended dose for the combination of HRS-1167 and famitinib. The latter phase II period is used to explore the efficacy of HRS-1167 plus famitinib /HRS-1167 plus famitinib plus camrelizumab as neoadjuvant therapy for gBRCA-mutated HER2-negative breast cancer. The primary endpoints in safety run-in period: the incidence of dose-limiting toxicity (DLT), the incidence and severity of adverse events (AE) and serious adverse events (SAE) ; in phase 2: the rate of pathological complete response (pCR) after surgery for each cohort as assessed by the investigator. Secondary endpoints included residual cancer burden (RCB) score, 3-year event-free survival (EFS), objective response rate (ORR), complete cell cycle arrest (CCCA) rate for HR+/HER2 - breast cancer, safety, and translational exploration study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 70 years old, female.
2. Patients with histologically confirmed unilateral primary invasive breast cancer who meet the criteria of cT0-4, N1-3, M0 or cT≥3, N0, M0 (inflammatory breast cancer not included).
3. Patients with HER-2 negative disease. HER2-negative disease was defined as follows: disease whose HER-2 is 1+ or negative by immunohistochemical (IHC), or fluorescence in situ hybridization (FISH) is negative if IHC is 2+.
4. Patients with pathogenic germline BRCA 1/2 mutation.
5. According to the RECIST 1.1 criteria, there is at least one measurable objective lesion.
6. Eastern Cooperative Oncology Group (ECOG) performance score 0-1.
7. Appropriate haematological, hepatic and renal function (no blood transfusion or hematopoietic stimulating factors within 14 days): 1) Absolute number of neutrophils (ANC) ≥ 1.5 x 10^9/L; 2) Platelets ≥ 100 x 10^9/L; 3) Hemoglobin ≥ 90 g/L ; 4) White blood cell (WBC) ≥ 3.0×10^9/L and ≤15×10^9/L; 5) Total bilirubin (TBIL) ≤ 1.5 times the upper limit of normal (ULN); 6) AST (SGOT) and ALT (SGPT) ≤ 2.5 x ULN; 7) serum creatinine (Cr) ≤1.5×ULN, and creatinine clearance (CrCL) ≥50 mL/min (Cockcroft-Gault equation); 8) Prothrombin time (PT) and activated partial thromboplastin time (APTT) ≤1.5 ULN with international normalized ratio (INR) ≤1.5 ULN (not receiving anticoagulation); 9) Serum albumin ≥ 2.5g/dL.
8. Left ventricular ejection fraction (LVEF) ≥ 50%.
9. 12-lead ECG: QT interval corrected by Fridericia method (QTcF) < 470 msec.
10. Urine test: urinary protein < 2+; If urinary protein ≥ 2+, 24-hour urinary protein quantification must show protein ≤1g.
11. Subject is willing and able to comply with the protocol (including contraceptive measures) for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
12. With good compliance with the planned treatment, are able to understand the follow-up procedures of this study and sigh the informed consent form.

Exclusion Criteria:

Patients with any of the following were not enrolled in the study:

1. Cancer-related history and treatment history: 1) Bilateral breast cancer; 2) Previous history of ductal carcinoma in situ (DCIS) or lobular carcinoma in situ (LCIS); 3) Previous history of invasive or metastatic breast cancer; 4) Any malignant tumor was diagnosed within 3 years before signing the informed consent, excluding cured cervical carcinoma in situ, basal cell carcinoma or squamous cell carcinoma; 5) Received systemic chemotherapy, systemic targeted therapy and local radiotherapy within 3 years before signing the informed consent; 6) Previously treated with VEGFR small molecule tyrosine kinase inhibitors (such as famitinib, sorafenib, sunitinib, regorafenib, etc.) (except bevacizumab); 7) Prior treatment with PARP inhibitors for any disease;
2. Stage IV breast cancer according to the AJCC staging system, 8th edition.
3. Inflammatory breast cancer or breast rupture.
4. There are clinical symptoms or diseases of the heart that are not well controlled
5. Hypertension that is not well controlled by antihypertensive medication: systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 90 mmHg has a history of hypertensive crisis or hypertensive encephalopathy.
6. NCI-CTCAE v5.0 grade ≥2 bleeding events occurred within 4 weeks before the first medication, including but not limited to hemoptysis (single episode of hemoptysis volume ≥ 2mL), vaginal bleeding, gastrointestinal bleeding, etc.
7. Excessive arterial/venous thrombosis events occurred within 6 months before the first medication, such as cerebrovascular accident (including transient ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism, etc. Patients with lower extremity intermuscular venous thrombosis who were evaluated as not requiring anticoagulant therapy, and those whose mural thrombus caused by catheterization had disappeared and did not require drug therapy were considered for enrollment.
8. Inability to swallow tablets normally or abnormal gastrointestinal function, which may affect drug absorption as judged by the researcher;
9. Receipt of a strong inhibitor of CYP3A4, CYP2D6, P-gp, or BCRP from the date of first dose <5 times of drug half-lives or 14 days; The interval between receiving treatment with the above enzyme strong inducers and the first dose < 28 days.
10. Evidence of any disease as judged by the investigator (e.g., severe or uncontrolled systemic disease, including severe systemic infection, uncontrolled hypertension, renal transplantation and active bleeding disease, coagulation disorders, platelet dysfunction, severe chronic gastrointestinal disease, or patients with other serious medical conditions);
11. Have undergone major surgery other than invasive diagnostic procedures, peripherally inserted central catheter (PICC) procedures, or pathological biopsy within 28 days prior to the first dose, or are expected to undergo major surgery during the study period;
12. Unhealed wounds, ulcers, or fractures;
13. Active hepatitis B (defined as hepatitis B surface antigen [HBsAg] positive and HBV-DNA ≥500IU/ml);
14. Hepatitis C infection (defined as a positive test for hepatitis C virus antibody [HCV-Ab] and an HCV-RNA test higher than the lower limit of the assay);
15. Known history of human immunodeficiency virus (HIV) infection;
16. Known history of psychotropic substance abuse, alcohol or drug abuse;
17. Active psychiatric disorders (schizophrenia, major depressive disorder, bipolar disorder, etc.) and depression being treated with antidepressants were not exclusion criteria.
18. Patients with known allergy or intolerance to the study drug or its excipents;
19. Patients of reproductive age who are pregnant or lactating, and who refuse to use appropriate contraception during the course of the trial;
20. Participated in other trial studies within 30 days before the first dose of the study drug, or not more than 5 half-lives since the last dose of the study drug;
21. Patients judged by the investigator to be ineligible for the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Safety run-in: Incidence rate of dose-limiting toxicities (DLTs) | 28±3 days
  Incidence rate of DLT will be evaluated in participants in the Safety Run-In, who will be followed for protocol-defined DLT events up to 28±3 days after the first dose of HRS-1167 and famitinib.
Safety run-in: adverse events (AEs) | 28±3 days
  Incidence rate of AEs of any cause will be evaluated in participants in the Safety Run-In according to CTCAE v5.0.
Safety run-in: Serious adverse events (SAEs) | 28±3 days
  Incidence rate of SAEs of any cause will be evaluated in participants in the Safety Run-In according to CTCAE v5.0.
Phase 2: Total Pathologic complete response (tpCR: ypT0/Tis ypN0) rate | Immediately after the surgery
  Defined as no residual invasive cancer cells are found in the pathological examination of breast and axillary lymph node; if only residual in situ cancer cells are present in the surgical specimens, it can also be considered as achieving a pathological complete response.

SECONDARY OUTCOMES:
Phase 2: Residual Cancer Burden (RCB) | Immediately after the surgery
  RCB will be estimated from routine pathological sections of the primary breast tumor site and the regional lymph nodes after the completion of neoadjuvant therapy. The pathological variables include bidimensional diameters of the primary tumor bed, the proportion of primary tumor area containing invasive carcinoma, the number of positive lymph nodes, and the diameter of the largest nodal metastasis
Phase 2: Event-free survival (EFS) | Approximately 3 years
  Defined as the time from the date of the first study dose to any of the following events: progression of disease that precludes surgery, local or distant recurrence, second primary malignancy (breast or other cancers) or death due to any cause.
Phase 2: Objective response rate (ORR) | Immediately after the surgery
  Defined as the proportion of patients with complete response (CR) and partial response (PR) by magnetic resonance imaging (MRI) according to RECIST v1.1.
Phase 2: Rate of complete cell cycle arrest (CCCA) in HR+/HER2- breast cancer | After 4 weeks of therapy
  Rate of CCCA determined by IHC Ki67 ( Ki67 ≤ 2.7%) between pre- and post-treatment.
Phase 2: Adverse events (AEs) | Up to 6 months
  Incidence rate of AEs of any cause will be evaluated in participants enrolled in the phase 2 period according to CTCAE v5.0.
Phase 2: Serious adverse events (SAEs) | Up to 6 months
  Incidence rate of SAEs of any cause will be evaluated in participants enrolled in the phase 2 period according to CTCAE v5.0.
Biomarker analysis1 | At baseline, at the end of first 2 cycles (each cycle is 28 days) and immediately after the surgery
  Gene mutations in the paired tumor and peripheral blood will be tested and analysed to predict therapy response.
Biomarker analysis 2 | At baseline, at the end of first 2 cycles (each cycle is 28 days) and immediately after the surgery
  Gene expression signatures in the paired tumor and peripheral blood will be tested and analysed to predict therapy response.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Ming Shao, MD, Principal Investigator — Fudan University
Locations (1):
- Breast cancer institute of Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided